CLINICAL TRIAL: NCT03824639
Title: Exercise Training to Improve Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E2545-P
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; exercise therapy; patient adherence
MeSH Terms: conditions — Cognitive Dysfunction; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Structured exercise
  Interventions: Behavioral: Structured exercise
- Control group (Active Comparator): Health education
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Structured exercise — Exercise instruction and encouragement
  Arms: Exercise group
Behavioral: Health Education — Provision of general information about a variety of health topics
  Arms: Control group

SUMMARY:
This project is assessing the feasibility of a novel home-based exercise intervention to improve episodic memory in individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
Background/Rationale:

Alzheimer's disease (AD) afflicts nearly 6 million Americans, a number projected to grow in coming decades. AD is known to have a long preclinical phase in which pathophysiologic processes develop many years, even decades, before the onset of clinical symptoms. During this preclinical phase there is evidence of unremitting decline in cognitive function, particularly in episodic memory. Thus far, evidence of the efficacy of pharmacological interventions to slow this decline in cognitive function has been limited, leading to increasing interest in the utility of nonpharmacological interventions including exercise.

Objective:

The investigators propose to assess the feasibility of a novel home-based exercise intervention to improve episodic memory in Veterans with mild cognitive impairment (MCI).

Methods:

The investigators will estimate the difference between the intervention (n=30) and the control group (n=30) on 6-month change in episodic memory (Rey-Osterrieth Complex Figure Test, Wechsler Logical Memory Test) as well as the effect size, which will be used as a basis for sample size calculation for a proposed larger study. Participants will be male and female Veterans 50 years of age or older with amnestic MCI.

ELIGIBILITY:
Inclusion Criteria:

* Amnestic MCI
* Ability to use a telephone without assistance

Exclusion Criteria:

* Angina Pectoris
* History of myocardial infarction within 6 months
* History of ventricular dysrhythmia requiring current therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Group | Control Group
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 25 | 27 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 27 | 29 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 31 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 26 | 30 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Wechsler Logical Memory Task [Mean (Standard Deviation); unit: units on a scale] — A recall test involving 2 short stories. Possible scores on the delayed recall task range from 0 (no details recalled for both stories) to 50 (all details recalled on both stories).
  units on a scale | 10.3 (5.6) | 9.5 (7.1) | 9.9 (6.4)
Rey-Osterrieth Complex Figure Test [Mean (Standard Deviation); unit: units on a scale] — A recall test involving a complex figure. Possible scores on the delayed recall task range from 0 (no accurate details recalled for the figure) to 36 (all details accurately recalled for the figure).
  units on a scale | 9.0 (4.6) | 7.6 (5.2) | 8.3 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Delayed Recall Score on Wechsler Logical Memory Task From Baseline to 6 Months
Description: Wechsler Logical Memory Task is a recall test involving 2 short stories. Possible scores on the delayed recall task range from 0 (no details recalled for both stories) to 50 (all details recalled on both stories). Outcome is change in the delayed recall score from baseline to 6 months.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 29 | 31
units on a scale | 0.74 (4.0) | -0.87 (4.7)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Other — Cohen's d will be used to estimate the effect size for comparing change in outcome measurements over 6 months in the exercise group to the control group. This effect size will be used for sample size calculations; Cohen's d = 0.37

2. Secondary Outcome: Change in Delayed Recall Score on the Rey-Osterrieth Complex Figure Test From Baseline to 6 Months
Description: Rey-Osterrieth Complex Figure Test is a recall test involving a complex figure. Possible scores on the delayed recall task range from 0 (no accurate details recalled for the figure) to 36 (all details accurately recalled for the figure). Outcome is change in the delayed recall score from baseline to 6 months.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 29 | 31
units on a scale | 1.18 (4.5) | 0.46 (3.3)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Cohen's d = 0.18

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03824639/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03824639/ICF_000.pdf